CLINICAL TRIAL: NCT04945083
Title: Gastrointestinal Tolerance and Acceptability of a High Protein, High Calorie Pudding in Adult Patients With/or at Risk for Malnutrition
Brief Title: Evaluation of a High Protein, High Calorie Pudding in Adults With/or at Risk for Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BL55
Record Dates: First submitted 2021-06-07; First posted 2021-06-30 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Gastrointestinal Tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Nutritional Pudding (Experimental): 2 servings per day
  Interventions: Other: Experimental Nutritional Pudding

INTERVENTIONS:
Other: Experimental Nutritional Pudding — High Calorie, High Protein pudding

SUMMARY:
This is a multi-center, prospective, non-randomized, non-blinded, single-arm, single treatment study to evaluate the tolerance of a nutritional pudding.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed and dated an ICF approved by an IEC, and provided applicable privacy authorization prior to any participation
* Subject is considered by a dietitian or clinician as malnourished or at risk for malnutrition based on current use of an oral nutritional supplement (ONS), recently identified as malnourished or at risk of malnutrition based on validated malnutrition screening tool or has had weight loss within last two months as a result of a hospitalization or chronic illness
* Subject currently has normal GI function
* Subject requires ONS and is willing to comply with the study protocol

Exclusion Criteria:

* Subject has severe dementia or delirium, eating disorder, history of significant neurological or psychiatric disorder affecting abilities to answer questions, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures
* Subject had a history of diabetes as evidenced by taking antihyperglycemic medications or by self-reported dietary modification
* Subject is currently taking or has taken antibiotics within 1 week prior to enrollment
* Subject has undergone major GI surgery less than 3 months prior to enrollment in the study
* Subject has current active malignant disease or was treated within the last 6 months for cancer, except basal or squamous cell skin carcinoma, prior to enrollment
* Subject has an immunodeficiency disorder
* Subject has had a myocardial infarction within the last 3 months prior to enrollment
* Subject is known to be allergic or intolerant to any ingredient found in the study product
* Subject has an aversion to any of the flavours of product being tested
* Subject has an obstruction of the GI tract precluding ingestion or absorption of the study product, inflammatory bowel disease, gastric esophageal reflux disease, short bowel syndrome, or other major gastrointestinal disease-causing symptoms including (but not limited to) uncontrollable severe diarrhea, nausea, or vomiting
* Subject is currently taking medications/dietary supplements/substances that could profoundly modulate metabolism or affect gastrointestinal motility
* Participation in another study that has not been approved as a concomitant study
* Subject has a clinical condition that is contraindicated with this product as determined by the clinician in accordance with standard of care
* Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Gastro-Intestinal Tolerance | Study Day 1 to Study Day 8
  Subject completed Bristol Stool Type questionnaire; Stool is classified into 7 groups (Types 1-7) with Type 3-4 as ideal stools

SECONDARY OUTCOMES:
Nutritional Supplement Palatability | Study Day 1 to Study Day 8
  Subject completed questionnaire; 4 questions scaled from 1 -Dislike Extremely to 9-Like Extremely; 2 questions scaled from Not at all Enough to Far Too
Nutritional Supplement Compliance | Study Day 1 to Study Day 28
  Subject completed daily intake questionnaire including amount of serving consumed

OTHER OUTCOMES:
Weight | Baseline to Study Day 28
  For BMI Calculation
Height | Baseline to Study Day 28
  For BMI Calculation
Medication Usage | Baseline to Study Day 28
  Subject reported medication usage
Adverse Events | Baseline to Study Day 28
  Subject reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Maria Camprubi, PhD, Study Chair — Abbott Nutrition
Locations (3):
- United Kingdom (3):
  - North Coast Medical Ltd, Newquay Health Centre, Newquay, Cornwall
  - The Alverton Practice, Atlantic Medical, Penzance, Cornwall
  - Morrab Surgery, Penzance, Cornwall

IPD SHARING:
Plan to Share IPD: No